CLINICAL TRIAL: NCT00736801
Title: Effect of Salmeterol on Brain-Derived Neurotrophic Factor (BDNF) Concentrations in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: PD Dr. med. Marek Lommatzsch, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LO-1111
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Allergic Asthma
Keywords: Airway hyperresponsiveness
MeSH Terms: conditions — Respiratory Hypersensitivity | interventions — Fluticasone-Salmeterol Drug Combination; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Treatment with Salmeterol for 2 weeks, followed by a treatment with Salmeterol and Fluticasone for 2 weeks.
  Interventions: Drug: Salmeterol and Salmeterol / Fluticasone

INTERVENTIONS:
Drug: Salmeterol and Salmeterol / Fluticasone — Patients inhale salmeterol for 2 weeks, followed by an inhalation of both salmeterol and fluticasone for 2 weeks.
  Other Names: Serevent; Viani

SUMMARY:
BDNF has been linked to the pathogenesis of airway hyperresponsiveness in asthma. In this trial, the impact of a treatment with salmeterol and salmeterol / fluticasone on BDNF concentrations will be assessed in patients with asthma. The investigators hypothesize that salmeterol impacts on BDNF concentrations in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, a physician's diagnosis of allergic asthma
* A documented sensitization to aero-allergens (pollen, animal hair, or house dust mite)
* A pre-bronchodilator forced expiratory volume in the first second (FEV1) > 80 % of the predicted value (% predicted), a provocative concentration of histamine causing a 20 % fall in FEV1 (PC20) of < 8 mg histamine / ml

Exclusion Criteria:

* No regular treatment (only short-acting inhalers on demand were allowed)
* No history of or evidence for any other chronic disease than asthma
* No history of smoking, absence of any signs or symptoms of an infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
BDNF concentrations in serum, platelets and plasma | 2006 - 2007

SECONDARY OUTCOMES:
Airway hyperresponsiveness | 2006 - 2007

CONTACTS AND LOCATIONS:
Overall Officials: Johann C. Virchow, MD, FCCP, Study Chair — University of Rostock
Locations (1):
- University of Rostock, Rostock, Germany

REFERENCES:
- [Background] Lommatzsch M, Schloetcke K, Klotz J, Schuhbaeck K, Zingler D, Zingler C, Schulte-Herbruggen O, Gill H, Schuff-Werner P, Virchow JC. Brain-derived neurotrophic factor in platelets and airflow limitation in asthma. Am J Respir Crit Care Med. 2005 Jan 15;171(2):115-20. doi: 10.1164/rccm.200406-758OC. Epub 2004 Oct 29. PMID 15516533
- [Derived] Lommatzsch M, Lindner Y, Edner A, Bratke K, Kuepper M, Virchow JC. Adverse effects of salmeterol in asthma: a neuronal perspective. Thorax. 2009 Sep;64(9):763-9. doi: 10.1136/thx.2008.110916. Epub 2009 Feb 22. PMID 19237390